CLINICAL TRIAL: NCT02688075
Title: Prospective, Observational, 12-month Assessment of Canagliflozin Treatment in Type 2 Diabetes Mellitus in a Usual Clinical Practice in Canada (CANadian CAnagliflozin REgistry: CanCARE)
Brief Title: An Observational Study to Assess the Canagliflozin Treatment in Type 2 Diabetes Mellitus in a Usual Clinical Practice in Canada
Acronym: CanCARE
Status: Completed | Type: Observational
Sponsor: Janssen Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR107542; 28431754DIA4012 (Other: Janssen Inc.)
Record Dates: First submitted 2016-02-17; First posted 2016-02-23 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus Type 2; Canagliflozin; Observational Study
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Canagliflozin Plus or Minus(+/-) Other Antihyperglycemic Agent: Participants who are receiving Canagliflozin +/- other antihyperglycemic agent (AHA) as per usual clinical practice will be observed for effectiveness, safety and PRO.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Participants who are receiving Canagliflozin +/- other AHA as per usual clinical practice will be observed for effectiveness, safety and PRO.

SUMMARY:
The purpose of this study is to evaluate canagliflozin use in the treatment of type 2 diabetes mellitus (T2DM) and generate evidence of its effectiveness, safety and patient-reported outcome (PRO) in a usual clinical practice in Canada.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, nation-wide, multicenter (more than one study site) study to evaluate the treatment of T2DM with canagliflozin in a usual clinical practice in Canada. Approximately 535 participants will be enrolled into this study. The planned study duration for each participant will be 12 months [plus or minus (+/-) 4 weeks], including 4 study visits in accordance with the usual clinical practice: enrollment and visits at 3, 6 and 12 months (+/- 4 weeks). Participants will primarily be observed for effectiveness, safety and PRO over an observational period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a diagnosis of type 2 diabetes mellitus (T2DM) with glycosylated hemoglobin (HbA1c) of greater than or equal to (>=) 7 percent (%) at baseline
* Participant must be on a stable antihyperglycemic treatment regimen for at least 30 days prior to canagliflozin initiation
* Participant must have estimated glomerular filtration rate (eGFR) >=60 milliliter (mL)/minute(min)/1.73 meter^2 (m^2)
* Must be a sodium-glucose co-transporter 2 (SGLT2) inhibitors naive participant initiating canagliflozin treatment prior to study enrollment
* Participant must provide a written consent for data collection by signing an ICF indicating that they understand the procedures for data collection and are willing to participate in the study

Exclusion Criteria:

* Participants with a history of SGLT2 inhibitors use (canagliflozin, empagliflozin, dapagliflozin or any other SGLT2 inhibitor)
* Participants with a history of diabetic ketoacidosis (DKA), autoimmune diabetes (example, type 1 diabetes mellitus [T1DM] and latent autoimmune diabetes in adults [LADA]), pancreas or beta-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy
* Participants who received an investigational drug (including vaccines) within 3 months before the initiation of canagliflozin
* Participant who is currently enrolled or plans to enroll in an investigational study
* Participant who is pregnant or breastfeeding or planning to become pregnant or breast feed during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry population will include Canadian sodium-glucose co-transporter 2 (SGLT2) naive type 2 diabetes mellitus (T2DM) participants, initiating canagliflozin as part of their optimal treatment approach, based on the independent clinical judgment of their treating physicians.
Sampling Method: Non-Probability Sample
Enrollment: 538 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Mean Glycosylated Hemoglobin (HbA1c) at 6 and 12 Months | Baseline, Month 6 and 12
  Mean HbA1c will be estimated.

SECONDARY OUTCOMES:
Change From Baseline in Mean Glycosylated Hemoglobin (HbA1c) at 3, 6 and 12 Months by HbA1c Subgroup | Baseline, Month 3, 6 and 12
  Mean HbA1c will be estimated.
Percentage of Participants Achieving Glycosylated Hemoglobin (HbA1c) Less Than (<) 7.0 Percent (%) | Month 3, 6 and 12
  Percentage of participants achieving HbA1c <7.0 will be evaluated.
Percentage of Participants Achieving Glycosylated Hemoglobin (HbA1c) Less Than (<) 6.5 Percent (%) | Month 3, 6 and 12
  Percentage of participants achieving HbA1c <6.5 will be evaluated.
Change From Baseline in Mean Weight at Month 3, 6 and 12 | Baseline, Month 3, 6 and 12
  Mean Weight will be estimated.
Change From Baseline in Body Mass Index (BMI) at Month 3, 6 and 12 | Baseline, Month 3, 6 and 12
  The BMI will be estimated.
Change From Baseline in Waist Circumference at Month 3, 6 and 12 | Baseline, Month 3, 6 and 12
  Waist Circumference will be estimated.
Percentage of Participants With Weight Loss From Baseline at Month 3, 6 and 12 | Baseline, Month 3, 6 and 12
  Percentage of participants with weight loss will be evaluated.
Percentage of Participants With Greater Than or Equal to (>=) 0.5% Reduction in Glycosylated Hemoglobin (HbA1c) Plus Weight Loss >=3% | Up to Month 12
  Percentage of participants with >= 0.5% reduction in HbA1c plus weight loss >=3% will be evaluated.
Current Health Satisfaction Questionnaire (CHES-Q) | Up to Month 12
  The responses to the questions of the CHES-Q and domain scores (physical, emotional, blood sugar, blood pressure and knowledge) will be evaluated.
Canagliflozin Treatment Adherence | Up to Month 12
  Treatment adherence will be based on percentage of prescribed pills taken in last 14 days as reported by participants.
Number of Participants with Adverse Events (AEs) and Serious AEs | Up to Month 12
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Inc. Clinical Trial, Study Director — Janssen Inc.
Locations (23):
- Canada (23):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Coquitlam, British Columbia
  - Surrey, British Columbia
  - Winnipeg, Manitoba
  - Brampton, Ontario
  - Downsview, Ontario
  - Guelph, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Ohsweken, Ontario
  - Ottawa, Ontario
  - Smiths Falls, Ontario
  - Toronto, Ontario
  - Laval, Quebec
  - Longueuil, Quebec
  - Montreal, Quebec
  - Saint-Jean-sur-Richelieu, Quebec
  - Saint-Marc-des-Carrieres, Quebec
  - Sherbrooke, Quebec
  - Toronto, Quebec
  - Westmont, Quebec
  - Saskatoon, Saskatchewan